CLINICAL TRIAL: NCT01959594
Title: Phase 1, Double Blind, Sponsor Open, Randomized, Placebo Controlled, Dose Escalation, Parallel Group Study To Investigate The Safety, Tolerability And Pharmacokinetics Of Repeat Doses Of PF-06412562 In Healthy Subjects
Brief Title: A Study To Observe Safety And Blood Concentrations Of PF-06412562 During And Following The Oral Administration Of Multiple Doses Of PF-06412562 In Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B7441002
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: multiple doses; pharmacokinetics; safety; tolerability; healthy volunteers; steady state; cognitive impairment associated with schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental)
  Interventions: Drug: 3 mg PF-06412562
- Cohort 2 (Experimental)
  Interventions: Drug: 10 mg PF-06412562
- Cohort 3 (Experimental)
  Interventions: Drug: 25 mg PF-06412562
- Optional Cohort 4 (Experimental)
  Interventions: Drug: PF-06412562 TBD mg
- Optional Cohort 5 (Experimental)
  Interventions: Drug: PF-06412562 TBD mg

INTERVENTIONS:
Drug: 3 mg PF-06412562 — oral dosing of 3 mg PF-06412562 tablets three times a day for 14 days
  Arms: Cohort 1
Drug: 10 mg PF-06412562 — oral dosing of 10 mg PF-06412562 tablets three times a day for 14 days
  Arms: Cohort 2
Drug: 25 mg PF-06412562 — oral dosing of 25 mg PF-06412562 tablets three times a day for 14 days
  Arms: Cohort 3
Drug: PF-06412562 TBD mg — oral dosing of PF-06412562 tablets three times a day for 14 days. Dosage and frequency to-be-determined based on previous cohorts
  Arms: Optional Cohort 4
Drug: PF-06412562 TBD mg — oral dosing of PF-06412562 tablets three times a day for 14 days. Dosage and frequency to-be-determined based on previous cohorts
  Arms: Optional Cohort 5

SUMMARY:
This study is designed to evaluate the safety and plasma concentrations of PF-06412562 in healthy volunteers following three times daily oral dosing of PF-06412562 for 14 days

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of non-childbearing potential and/or male subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs);

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Safety and toleration assessed by: adverse events, supine and standing vital sign measurements, electrocardiogram (ECG) standard 12 lead, blood and urine safety laboratory tests ,CogState and C-SSRS. | 0-15 days
Pharmacokinetics: Cmax, Tmax, AUCτ Ctrough, PTR, Rac on Cmax and AUCτ t1/2, CL/F, PTR, | 0-15 days
CogState at followup | 22-25 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7441002&StudyName=A%20Study%20To%20Observe%20Safety%20And%20Blood%20Concentrations%20Of%20PF-06412562%20During%20And%20Following%20The%20Oral%20Administration%20Of%20Multiple%20Doses%20Of%20PF